CLINICAL TRIAL: NCT05946837
Title: Near-infrared Fluorescence Lymphatic Imaging Assessment of Lymphatic Response to Pneumatic Back/Neck Lymphatic Drainage Delivered by a Pneumatic Manual Lymphatic Drainage Device
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Eva MedTech, Inc. (Unknown)
Responsible Party: Principal Investigator, Melissa B Aldrich, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-23-0093
Record Dates: First submitted 2023-06-29; First posted 2023-07-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Neck Pain; Back Pain
MeSH Terms: conditions — Neck Pain; Back Pain | interventions — Indocyanine Green; Coloring Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Pneumatic Compression Therapy (PCT) (Experimental)
  Interventions: Drug: Indocyanine green (ICG) dye; Device: NIRF-LI imaging; Device: Neuroglide pad

INTERVENTIONS:
Drug: Indocyanine green (ICG) dye — ICG (25 mg vial) will be reconstituted with 10 ml sterile water provided by the manufacturer; further dilutions will be made in sterile saline just prior to administration. The final concentration of 0.32 millimolar (mM) will provide 25 μg ICG/injection, with each injection of 0.1 cc to be made . Up to 30 intradermal injections using conventional 30- or 31-gauge needles will be administered to each subject, for a maximum dose of 750 ug ICG, over 200 times less than the maximum allowed dose. Injection sites will be cleaned with alcohol wipes before intradermal injection.
Device: NIRF-LI imaging — Near-infrared fluorescence lymphatic imaging (NIRF-LI) imaging will be done to assess the drainage of ICG laden lymph from ICG injection sites toward regional nodal basins for 60 minutes before, during and after the Neuroglide pad treatment
Device: Neuroglide pad — After injection of Indocyanine green (ICG) dye and NIRF-LI imaging the subject will lie on the Neuroglide pad for the one-hour PCT treatment session.

SUMMARY:
The purpose of this study is to objectively assess lymphatic function before, during, and immediately after Neuroglide treatment in lower trunk and leg lymphatic vessels, torso, axillary regions, inguinal regions, upper extremities, and cervical/neck and to determine any VAS (Visual Analog Scale, a commonly used measure of pain perception) score change after Neuroglide treatment.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory and possess all four limbs
* Female participants of childbearing potential must have a negative urine pregnancy test within 36 hours prior to study drug administration
* Female participants of childbearing potential must agree to use a medically accepted method of contraception for a period of one month following each imaging session in the study
* Weight less than 400 lbs

Exclusion Criteria:

* Women who are pregnant or breast-feeding
* Persons who are allergic to iodine or indocyanine green
* Heart failure, poorly controlled kidney disease (glomerular filtration rate <30 mls per minute), hypoproteinemia, pulmonary hypertension, or hypothyroidism
* Any circumstance where increased lymphatic or venous return is undesirable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-08-29 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Change in frequency of lymphatic pulsing as assessed by the number of lymphatic pulses per minute in each region imaged | Baseline, during Neuroglide treatment ( 1 hour after NIRF-LI imaging ), 1 hour after PCT treatment

SECONDARY OUTCOMES:
Change in pain as assessed by the Visual Analog Scale (VAS) | Baseline, 1 hour after PCT treatment, 4-8 weeks after imaging for data analysis completion
  This is scored from 1(no pain)-10( worst pain possible) a higher number indicating more pain

CONTACTS AND LOCATIONS:
Overall Officials: Melissa B Aldrich, PhD, MBA, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No